CLINICAL TRIAL: NCT03337464
Title: The Effects of a Single Bout of Exercise in Parkinson's Disease.
Brief Title: Single Exercise Bout in Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Parkinson's Research Centre (Other)
Responsible Party: Principal Investigator, A. Jon Stoessl, Clinical Director of PET, Pacific Parkinson's Research Centre
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-00084
Record Dates: First submitted 2017-02-18; First posted 2017-11-09 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: exercise; EEG; EMG; Motor function; Mood; Cognition
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1 PD group and 1 one age matched non-PD subjects
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to subject group and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease (Experimental): Subjects with Parkinson's disease
  Interventions: Other: cycling exercise
- Control (Active Comparator): Subjects without Parkinson's disease
  Interventions: Other: cycling exercise

INTERVENTIONS:
Other: cycling exercise — 5 x 3 minute bouts of cycling exercise separated by 3 minute rest periods

SUMMARY:
To assess 30 active people (15 with PD, 15 without) before and after 30 minutes of pedaling exercise using EEG-EMG, cognitive, mood and motor assessments.

DETAILED DESCRIPTION:
Purpose: To assess 15 subjects with PD and 15 healthy controls, who exercise on a regular basis, before, during and after 30 minutes of pedaling exercise intervention. The investigators will assess subjects for alterations in motor cortex assessment, cognition and mood as measured by EMG/EEG, motor assessment and several batteries of questionnaires. Findings from this study will lay the foundation for long-term studies.

Hypotheses: The investigators anticipate to observe an altered involvement of motor cortex during steady pedaling in individuals suffering from PD. In healthy control subjects it is anticipated that changes in cognition will be observable.

Justification: Hindered movement initiation and continuing locomotion is a common syndrome in PD with profound impact on the patient's mobility and quality of life. So far, the underlying pathophysiology is not completely understood. Since the observation that cortical activity contributes to the muscle activity during locomotion-like tasks underpins the importance of corticospinal function in humans, it is of importance to examine whether this cortical involvement is altered and displays abnormalities in patients with PD. Thus, the approach of corticomuscular coupling during a locomotion-like task would allow for better understanding of the pathophysiology of PD, a prerequisite to develop therapies. Findings of this study will lay the foundation for future long-term studies.

Additionally, by examining the oscillatory EEG patterns during the exercise intervention, the investigator will be able to read out the dose response curve in real time, which will provide information on the optimum intensity and duration of exercise. Findings will help to design future studies and to develop efficient exercise therapy interventions for people with PD.

People living with PD often suffer from cognitive decline, depression, and fatigue. By assessing cognitive function before and after the exercise intervention, there will be laid a foundation for future studies investigating the effect of exercise on cognition. The collected pilot data will be relevant to learn more about the effects of exercise on mood and fatigue as well as concomitant obstacles and facilitators during exercise interventions in patients with PD.

Objectives: The primary objective of this study is to investigate if activity that arises in the motor cortex and contributes to the muscle activity during moderate pedaling is altered in patients with PD compared to healthy gender- and age-matched controls. Thus, to better understand the role of the motor cortex and its contribution in simple automated repetitive tasks in patients with PD there will be analysis of the coherence of the coupling between EEG and EMG from active leg muscles during cycling on a stationary bicycle both in subjects with PD and age and gender matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 40-80 years
* Hoehn and Yahr stage I-III
* Exercise on a regular basis (at least 100 minutes of aerobic exercise per week)
* Montreal Cognitive Assessment score >/= 24
* Able to communicate with study personnel
* Able to be informed of the nature of the study and willing to give written consent form

Exclusion Criteria:

* Hoehn and Yahr stages IV-V
* Significant cardiovascular disease
* Previous stroke
* Not exercising on a regular basis
* Functional disabling dyskinesia
* Functional disabling dystonia
* Smoker
* Significant neurological or psychiatric illness other than PD
* Dementia
* Severe depression
* Significant musculoskeletal disorder (e.g. arthritis)
* Significant metabolic disorder (e.g. diabetes)
* Brain surgery in the past
* Currently taking beta blocker medication

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
EEG-EMG coherence | The change from immediately before, during, and immediatly after the single bout of exercise.
  Coherence of the coupling between EEG and EMG from active leg muscles during cycling on a stationary bicycle both in subjects with PD and age and gender matched healthy controls.

SECONDARY OUTCOMES:
Motor function | Immediately before and after the single bout of exercise.
  Examine motor function with the Movement disorders society unified Parkinson's disease rating scale motor section (MDS-UPDRS III)
Motor function | Immediately before and after the single bout of exercise.
  Examine motor function with the finger tapping
Motor function | Immediately before and after the single bout of exercise.
  Examine motor function with the Purdue pegboard
Motor function | Immediately before and after the single bout of exercise.
  Examine motor function with the Timed-up-and-go (TUG)
Cognitive function | Immediately before, after and at 3 hours following the single bout of exercise.
  Examine cognitive function with Montreal cognitive assessment (MoCA)
Cognitive function | Immediately before, after and at 3 hours following the single bout of exercise.
  Examine cognitive function with Verbal fluency
Cognitive function | Immediately before, after and at 3 hours following the single bout of exercise.
  Examine cognitive function with trail making test (A and B) and reaction time
Mood function | Immediately before, after and at 3 hours following the single bout of exercise.
  Examine mood with the Positive and Negative Affect Schedule.
Mood function | Immediately before, after and at 3 hours following the single bout of exercise.
  Examine mood with the Starkein Apathy scale

CONTACTS AND LOCATIONS:
Overall Officials: Silke Cresswell, MD, Principal Investigator — Pacific Parkinson's Research Centre
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No